CLINICAL TRIAL: NCT03864874
Title: Thoracoscopic Ultrasonography Versus Manual Lung Palpation by Thoracotomy for the Identification of Lung Nodules During Pulmonary Metastasectomy. A Prospective Blinded Cross-over Trial.
Brief Title: Use of Thoracoscopic Intraoperative Lung Ultrasound to Identify Pulmonary Metastases in Patients Submitted to Pulmonary Metastasectomy With Radical Intent.
Acronym: VATS-US1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Principal Investigator, Francesco Londero, Principal Investigator, Azienda Sanitaria-Universitaria Integrata di Udine
Other Study IDs: 30948
Record Dates: First submitted 2019-02-22; First posted 2019-03-06 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Pulmonary Metastases
Keywords: Pulmonary metastases; Intraoperative ultrasonography; Thoracoscopy; Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Intraoperative intracavitary lung ultrasonography — Ultrasonography on the deflated lung for detection of lung nodules

SUMMARY:
Experience drawn from many scientific articles showed that many patients who develop a limited pattern of pulmonary metastases after treatment of a primary tumor may benefit from surgical resection of the lung deposits. Pulmonary metastasectomy with curative intent is widely performed with the aim of prolonging life and, in some cases, being curative. Usually the surgical strategy is defined based on analysis of radiological investigations, performed during a follow-up program after resection of a tumor. However, many studies showed that the actual sensitivity of this examinations, namely computed tomography (CT) and positron-emission tomography (PET) is far from being 100% and finding further unexpected nodules at operation with lung manual palpation is not uncommon. Many surgeons perform pulmonary metastasectomy with a minimally invasive approach, in view of a less morbid and more cosmetic approach, but lung palpation is considerably hampered and surgical radicality might be impaired. With this study the investigators want to assess the ability of lung ultrasonography performed via a key-hole access (thoracoscopy, VATS) in detecting lung nodules compared with the standard practice represented by open thoracotomy, that is a wider incision that allows manual exploration of the organ. Therefore, every patient enrolled will undergo a double phase surgical approach: a first phase by thoracoscopy where a thorough lung ultrasonography will be performed and number and position of lung nodules will be annotated, and a second phase by open thoracotomy where lung is palpated and suspicious nodules will be removed. The incisions used for the first phase will be extended for the second, rendering any other procedure for the execution of lung ultrasonography unnecessary.

Should this study demonstrate a non-inferiority of lung ultrasonography in detecting lung nodules compared with manual palpation of the lung, patients should be offered a less invasive approach for treatment of their condition with no concerns regarding a potential lower therapeutic effect.

DETAILED DESCRIPTION:
Pulmonary metastasectomy is a surgical practice that poses many aspects of debate: standard approach has historically been represented by open thoracotomy, but video-assisted thoracic surgery (VATS) became an appealing alternative due to the lower surgical impact on the patient. Some authors blame the minimally invasive approach for pulmonary metastasectomy as less effective from an oncologic point of view since lung palpation is hampered, leading to reduced ability to identify unexpected nodules and potential impairment of surgical radicality.

Indeed, several papers demonstrated a suboptimal sensitivity of computed tomography (CT) and positron-emission tomography (PET) in detecting lung metastases and discover of further unexpected nodules at thoracotomy are not an uncommon eventuality.

A few authors demonstrated the utility of intraoperative lung ultrasound performed through a VATS approach (VATS-US) in identifying lung nodules. However, the real effectiveness of this technique has never been prospectively compared with the current gold standard represented by open thoracotomy and lung manual exploration. Aim of our study is to assess the non-inferiority of VATS-US compared with manual palpation to identify lung nodules during pulmonary metastasectomy.

The study design is a monocentric non-inferiority diagnostic crossover trial, based on the execution of intraoperative lung ultrasound (VATS-US) in patients undergoing pulmonary metastasectomy with radical intent. Aim of the study is to assess the non-inferiority of the ultrasonographic investigation on the lung parenchyma performed via a thoracoscopic approach in identifying lung nodules compared with manual organ palpation by thoracotomy.

Study design After general anesthesia administration patients will be intubated with a double lumen tube and positioned in a standard lateral decubitus. Thereby the target lung will be excluded from ventilation and deflated. After creation of 2-3 thoracoscopic ports the lung is explored under thoracoscopic vision with a laparoscopic ultrasound probe (Esaote LP323, Esaote, Genova, Italy) by a surgeon with experience on the use of lung ultrasound. Data regarding number, size, depth and lobar localization of nodules are registered on a data collection paper. The surgeon who performed the investigation therefore leaves the operative room and another surgeon, blind to the previous phase findings, performs an anterolateral thoracotomy and an accurate palpation of the lung. Suspicious nodules are therefore resected and sent for histology. Data on number and localization of excised nodules are registered on a separate collection paper. Results from both phases are then compared and matched with histology report.

Thoracotomy will be performed extending the length of the utility port. The others 1-2 hole are eventually used for insertion of chest drainage tubes, that in our institution are routinely positioned following any intervention within the pleural space. Consequently, no adjunctive incision will be performed for the execution of VATS-US compared with a standard thoracotomy approach. Only after nodules resection the two surgeons will compare their findings in order to make sure that any nodule identified at VATS-US but not at thoracotomy has not been omitted. The execution of the ultrasonographic investigation will require an appropriate lung deflation. Therefore, in some cases air aspiration from the target lung with a small catheter inserted through the endobronchial tube will be required, as previously described in other studies.

In order to guarantee patients' safety, they will never be left unattended during all phases of the intervention, and execution of any required urgent procedure for rare intraoperative complications will never be delayed, including those that may interfere with the execution of the ultrasonographic exam. It has been calculated that operative time will be extended of about 20-30 minutes to allow the execution of VATS-US.

No extra procedure or drugs administration will be required for the study. Only nodules that will be considered suspicious by the second surgeon during the thoracotomic phase or after discussion between the two operators will be excised, as expected in the standard practice.

The investigators will collect data regarding patients' features (age, biometric measurements, preoperative lung function tests data, lung comorbidities), preoperative CT scan findings (number, size and localization of lung nodules), ultrasonographic findings (number, size, depth, localization and shape of lung nodules), number and localization of nodules excised at thoracotomy, histology report data (histological nature, size, depth of lung nodules), time of surgery and of VATS-US, incidence of post-operative adverse events.

Sample size and statistical analysis Sensitivity and specificity of VATS-US will be calculated compared with manual palpation. The inter-rater agreement will be measured by calculating Cohen's kappa coefficient. Continuous data will be summarized as mean and standard deviation or median and twenty-fifth to seventy-fifth percentiles in case of non-normal distributions. Normality will be assessed by using Shapiro-Wilk test. Categorical variables will be reported as counts and percentages. Comparisons will be carried out using paired t-test, Wilcoxon signed ranks test and McNemar test where appropriate.

STATA software (release 14 StataCorp LP, College Station, TX, USA) will be utilized for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient candidate to pulmonary metastasectomy with curative intent by mean of both major anatomical or limited resection;
* Age > 18 years.

Exclusion Criteria:

* Patients with widespread metastatic disease where surgical resection is performed only for diagnostic purposes;
* History of previous intrapleural talc injection;
* Any anatomical or pathological condition (eg. diffuse adhesions, severe emphysema) that may interfere with execution of ultrasonographic investigation;
* Incomplete lung exclusion during surgical procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with pulmonary oligometastases from various primary cancers.
Sampling Method: Probability Sample
Enrollment: 89 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of nodules/lesions identified: surgery | Intraoperative
  Number of nodules identified at VATS-US and lung palpation/ number of lesions identified at lung palpation
Number of nodules/lesions identified: histology | Up to 2 weeks
  Number of nodules identified at VATS-US and lung palpation/ number of lesions confirmed to be pulmonary metastases

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Londero, MD, Principal Investigator — Thoracic Surgery Unit, ASUI S Maria della Misericordia, Udine; Angelo Morelli, MD, Study Director — Thoracic Surgery Unit, ASUI S Maria della Misericordia, Udine; Sandro Gelsomino, MD, PhD, FESC, Study Chair — Cardiothoracic Department Maastricht University Hospital, Maastricht, The Netherlands; Luigi Castriotta, MD, Study Chair — Clinical Epidemiology Department, ASUI S Maria della Misericordia, Udine; William Grossi, MD, Study Chair — Thoracic Surgery Unit, ASUI S Maria della Misericordia, Udine; Gianluca Masullo, MD, Study Chair — Thoracic Surgery Unit, ASUI S Maria della Misericordia, Udine
Locations (1):
- Thoracic Surgery Unit, Cardiothoracic Dept., ASUI S Maria della Misericordia, Udine, Ud, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Molnar TF, Gebitekin C, Turna A. What are the considerations in the surgical approach in pulmonary metastasectomy? J Thorac Oncol. 2010 Jun;5(6 Suppl 2):S140-4. doi: 10.1097/JTO.0b013e3181dcf62c. PMID 20502249
- [Background] Ellis MC, Hessman CJ, Weerasinghe R, Schipper PH, Vetto JT. Comparison of pulmonary nodule detection rates between preoperative CT imaging and intraoperative lung palpation. Am J Surg. 2011 May;201(5):619-22. doi: 10.1016/j.amjsurg.2011.01.005. PMID 21545910
- [Background] Eckardt J, Licht PB. Thoracoscopic or open surgery for pulmonary metastasectomy: an observer blinded study. Ann Thorac Surg. 2014 Aug;98(2):466-9; discussion 469-70. doi: 10.1016/j.athoracsur.2014.04.063. Epub 2014 Jun 11. PMID 24928676
- [Background] Macherey S, Doerr F, Heldwein M, Hekmat K. Is manual palpation of the lung necessary in patients undergoing pulmonary metastasectomy? Interact Cardiovasc Thorac Surg. 2016 Mar;22(3):351-9. doi: 10.1093/icvts/ivv337. Epub 2015 Dec 17. PMID 26678151
- [Background] Piolanti M, Coppola F, Papa S, Pilotti V, Mattioli S, Gavelli G. Ultrasonographic localization of occult pulmonary nodules during video-assisted thoracic surgery. Eur Radiol. 2003 Oct;13(10):2358-64. doi: 10.1007/s00330-003-1916-6. Epub 2003 May 8. PMID 12736756
- [Background] Rocco G, Cicalese M, La Manna C, La Rocca A, Martucci N, Salvi R. Ultrasonographic identification of peripheral pulmonary nodules through uniportal video-assisted thoracic surgery. Ann Thorac Surg. 2011 Sep;92(3):1099-101. doi: 10.1016/j.athoracsur.2011.03.030. PMID 21871306
- [Background] Mattioli S, D'Ovidio F, Daddi N, Ferruzzi L, Pilotti V, Ruffato A, Bolzani R, Gavelli G. Transthoracic endosonography for the intraoperative localization of lung nodules. Ann Thorac Surg. 2005 Feb;79(2):443-9; discussion 443-9. doi: 10.1016/j.athoracsur.2004.07.087. PMID 15680811
- [Background] Pastorino U, Buyse M, Friedel G, Ginsberg RJ, Girard P, Goldstraw P, Johnston M, McCormack P, Pass H, Putnam JB Jr; International Registry of Lung Metastases. Long-term results of lung metastasectomy: prognostic analyses based on 5206 cases. J Thorac Cardiovasc Surg. 1997 Jan;113(1):37-49. doi: 10.1016/s0022-5223(97)70397-0. PMID 9011700
- [Background] Vannucci F, Gonzalez-Rivas D. Is VATS lobectomy standard of care for operable non-small cell lung cancer? Lung Cancer. 2016 Oct;100:114-119. doi: 10.1016/j.lungcan.2016.08.004. Epub 2016 Aug 11. PMID 27597290
- [Background] Internullo E, Cassivi SD, Van Raemdonck D, Friedel G, Treasure T; ESTS Pulmonary Metastasectomy Working Group. Pulmonary metastasectomy: a survey of current practice amongst members of the European Society of Thoracic Surgeons. J Thorac Oncol. 2008 Nov;3(11):1257-66. doi: 10.1097/JTO.0b013e31818bd9da. PMID 18978560
- [Background] Lobo V, Weingrow D, Perera P, Williams SR, Gharahbaghian L. Thoracic ultrasonography. Crit Care Clin. 2014 Jan;30(1):93-117, v-vi. doi: 10.1016/j.ccc.2013.08.002. PMID 24295842
- [Background] Ujiie H, Kato T, Hu HP, Hasan S, Patel P, Wada H, Lee D, Fujino K, Hwang DM, Cypel M, de Perrot M, Pierre A, Darling G, Waddell TK, Keshavjee S, Yasufuku K. Evaluation of a New Ultrasound Thoracoscope for Localization of Lung Nodules in Ex Vivo Human Lungs. Ann Thorac Surg. 2017 Mar;103(3):926-934. doi: 10.1016/j.athoracsur.2016.08.031. Epub 2016 Oct 17. PMID 27765176
- [Background] Gossot D, Radu C, Girard P, Le Cesne A, Bonvalot S, Boudaya MS, Validire P, Magdeleinat P. Resection of pulmonary metastases from sarcoma: can some patients benefit from a less invasive approach? Ann Thorac Surg. 2009 Jan;87(1):238-43. doi: 10.1016/j.athoracsur.2008.09.036. PMID 19101304
- [Derived] Londero F, Castriotta L, Grossi W, Masullo G, Morelli A, Tetta C, Livi U, Maessen JG, Gelsomino S. VATS-US1: Thoracoscopic ultrasonography for the identification of nodules during lung metastasectomy. Future Oncol. 2020 Feb;16(5):85-89. doi: 10.2217/fon-2019-0608. Epub 2020 Jan 9. PMID 31916464